CLINICAL TRIAL: NCT05614947
Title: Impact of 60 Days Powdered Tart Cherry Supplementation on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor of Exercise Physiology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-F-16
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tart cherry (Experimental): two capsules daily for 60 days
  Interventions: Dietary Supplement: Powdered tart cherry
- placebo (Placebo Comparator): two capsules daily for 60 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Powdered tart cherry — 500 mg freeze-dried tart cherry per capsule
  Arms: tart cherry
Dietary Supplement: Placebo — 500 mg colored cornstarch per capsule
  Arms: placebo

SUMMARY:
Metabolic syndrome (MetSyn) is a growing health concern, with up to 25% of the worlds population having the syndrome. MetSyn is a primary risk factor for cardiovascular disease and type II diabetes development, and is independently associated with all-cause mortality, making it an important disease target. The primary treatment for MetSyn is exercise and weight loss, along with medically necessary treatment. Exercise, along with dietary changes such as increased fiber and polyphenol intake can positively impact many of the metabolic abnormalities seen with MetSyn. For example, polyphenols have been shown to decrease lipid concentration and improved glucose clearance as well as decreased oxidative stress and inflammation. Powdered tart cherry capsules, which contain the skin of the fruit, provides polysaccharides (fiber) that would likely act as a substrate for gut bacteria degradation, providing energy substrates and barrier integrity to the colonocytes and increasing the bioavailability of the polyphenols to other cells in the body. However there have been no long-term investigations into the use of powdered tart cherry supplements in MetSyn, therefore we aim to determine if 60 days tart cherry supplementation modify criteria for MetSyn in currently diagnosed individuals including body mass, waist circumference, blood pressure, blood lipid levels and blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with metabolic syndrome by a physician or meet the diagnostic criteria: Waist circumference greater than 40 inches (men) or greater than 35 inches (women), High blood pressure (greater than 130/80) or taking medication for high blood pressure, High triglycerides (greater than 150 mg/dL) or low HDL (less than 40 for men, less than 50 for women), High fasting blood glucose (100-126 mg/dL) or diagnosed as pre-diabetic
* Age 25-60

Exclusion Criteria:

* currently taking medication for glucose or lipid control, such as metformin and/or statin
* currently using anti-inflammatory medications & have not used corticosteroids in the last two months
* diagnosed with or currently being treated for an inflammatory condition
* major organ system impairment (heart failure, renal failure, severe impairment of respiratory function)
* currently a smoker or quit less than 12 months ago

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Change in baseline systolic and diastolic blood pressure | baseline, 60 days post supplmentation
Change in fasting high-density lipoprotein (HDL) cholesterol | baseline, 30 days post supplementation, 60 days post supplmentation
Change in fasting triglyceride levels | baseline, 30 days post supplementation, 60 days post supplmentation
Change in fasting blood glucose level | baseline, 30 days post supplementation, 60 days post supplmentation
Change in waist circumference | baseline, 60 days post supplmentation
Change in body fat distribution | baseline, 60 days post supplmentation
Change in erythrocyte sedimentation rate | baseline, 30 days post supplementation, 60 days post supplmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No